CLINICAL TRIAL: NCT06678126
Title: Randomized Phase II 2 by 2 Factorial Trial of Adaptive Versus Non-adaptive Radiotherapy and 2 Bladder Filling Instructions for Patients with Intermediate or High Risk Localized Prostate Cancer (ARP)
Brief Title: Adaptive Versus Non-adaptive Radiotherapy and 2 Bladder Filling Instructions for Patients with Intermediate or High Risk Localized Prostate Cancer (ARP)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Scott Tyldesley (Other)
Responsible Party: Sponsor-Investigator, Scott Tyldesley, MD MPA ABR FRCPC, British Columbia Cancer Agency
Organization: British Columbia Cancer Agency (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: ARP
Record Dates: First submitted 2024-11-04; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer
Keywords: adaptive radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized Phase II 2 by 2 factorial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1i (Active Comparator): Adaptive RT & Standard Bladder Filling Instructions
  Interventions: Radiation: Prostate and Pelvic Nodes Radiotherapy
- Arm 1ii (Active Comparator): Adaptive RT and Custom Bladder Filling Instructions
  Interventions: Radiation: Prostate and Pelvic Nodes Radiotherapy
- Arm 2i (Active Comparator): Non Adaptive RT and Standard Bladder Filling Instructions
  Interventions: Radiation: Prostate and Pelvic Nodes Radiotherapy
- Arm 2ii (Active Comparator): Non Adaptive RT and Custom Bladder Filling Instructions
  Interventions: Radiation: Prostate and Pelvic Nodes Radiotherapy

INTERVENTIONS:
Radiation: Prostate and Pelvic Nodes Radiotherapy — 60 Gy prostate and 44 Gy pelvic nodes with 20 fractions

SUMMARY:
The study is being done to compare the side effects between two different radiation techniques, standard non-adaptive radiation therapy vs. daily adaptive radiation therapy and also comparing two different bladder filling instructions to find out if customized bladder instructions may lead to better treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Pathological diagnosis of a primary prostate adenocarcinoma
* NCCN Intermediate or high risk localized prostate cancer and clinically N0 and M0 by conventional imaging
* Intermediate: one or more of cT2b-T2c, PSA 10-20, or Gleason Group 2 or 3

  * High: one or more of: cT3a, PSA > 20, or Gleason Group 4 or 5.
  * Consented to RT with moderate hypofractionated RT to pelvic nodes (44 Gy) and prostate (60Gy) in 20 fractions using standard BC Cancer regimen
* Able to complete BC Cancer POSI questionnairesWilling to attend adaptive treatment slot timing as required by treating centre.
* Willing and able to have regular per protocol follow up and blood work
* Feasible to start protocol treatment within 120 calendar days of participant enrolment
* Continent of urine (or able to maintain continence with penile clamp/cuff during RT as needed) and able to follow bladder filling instructions.
* Baseline IPSS score < 20 at time of enrolment.
* ECOG performance Status : 0-2.
* Nodal risk ≥ 20% using the Memorial Sloan Kettering Nodal Risk Nomogram (https://www.mskcc.org/nomograms/prostate/pre_op).
* Negative for bone metastases on bone scan within 3 months of enrolment
* No involved nodes on Abdomen and pelvic CT or pelvic MRI within 3 months of enrolment.

Exclusion Criteria:

* Indwelling urinary catheter.
* Hip prosthesis
* Prior pelvic radiotherapy
* Unable to lie still on RT treatment couch for more than 30 minutes
* Clinical T3b or T4 tumours
* Prior transurethral resection of prostate or radical prostatectomy
* Presence of a pelvic kidney.
* Prior pelvic radiotherapy.
* Significant urinary incontinence: ie > 1 soaked, or 2 non-soaked pads per day.
* Inflammatory bowel disease, systemic lupus erythematosis, scleroderma, or other connective tissue disorders other than rheumatoid arthritis.
* Metastatic disease identified on staging investigations.
* Any other serious intercurrent illness or medical condition judged by the local investigator to compromise the participant's safety, preclude safe administration of the planned protocol treatment, or prevent the participant from being managed according to the protocol guidelines
* Potentially fertile patient who are unwilling to employ highly effective contraception

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2033-06 (Estimated); Study Completion 2035-01 (Estimated)

PRIMARY OUTCOMES:
Assess the feasibility of randomization to adaptive vs standard radiotherapy localized high-risk prostate cancer. | Accrual period, estimated 3.5 years
  Accrual and randomization rate will be captured in REDCap database until the goal of 104 participants are randomized. With the accrual rate, we may imply it is feasible to do a larger more definitive and timely randomized control trial.

SECONDARY OUTCOMES:
Measure and compare the patient reported Acute GU and GI bladder toxicity associated standard (SRT) and Adaptive (ART) radiotherapy for localized prostate cancer. | 5 years after participant completes RT
  using Patient reported questionnaire (POSI) to review toxicities at 1.5 months, 6 months, and years 1,2,5 post study RT.
Measure and compare the patient reported Late GU and GI bladder side effects associated standard (SRT) and Adaptive (ART) radiotherapy for localized prostate cancer. | 5 years after participant completes RT
  using Patient reported questionnaire (POSI) to review toxicities at 1.5 months, 6 months, and years 1,2,5 post study RT.
Measure and compare the physician reported CTCAE Acute (6 weeks post RT) GU and GI bladder CTCAE toxicity associated standard (SRT) and Adaptive (ART) radiotherapy for localized prostate cancer | 5 years after participant completes RT
  review toxicities at 1.5 months, 6 months, and years 1,2,5 post study RT.
Determine which bladder filling instructions (BFI) are associated with daily shortest treatment time | approx 4 weeks during treatment of 20 fractions
  using treatment time record during the 20 fractions
Determine which BFIs are associated with least rescan and repeat CBCT requirements | approx 4 weeks during treatment of 20 fractions
  using records from treatment

CONTACTS AND LOCATIONS:
Locations (1):
- BC Cancer Vancouver, Vancouver, British Columbia, Canada